CLINICAL TRIAL: NCT02397694
Title: A Phase 2, Randomized, Double-Blinded Study of the Safety and Efficacy of GS-9883 + Emtricitabine/Tenofovir Alafenamide Versus Dolutegravir + Emtricitabine/Tenofovir Alafenamide in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Brief Title: Safety and Efficacy of Bictegravir + Emtricitabine/Tenofovir Alafenamide Versus Dolutegravir + Emtricitabine/Tenofovir Alafenamide in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-141-1475
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: HIV-1 Infection
Keywords: Adult; HIV; naive
MeSH Terms: interventions — imidazole mustard; bictegravir; dolutegravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BIC + F/TAF (Experimental): Participants will receive BIC + F/TAF FDC + DTG placebo for 48 weeks.
  * Following Week 48, participants will continue to take their blinded treatment and attend visits every 12 weeks until treatment assignments have been unblinded. Participants will return for an unblinding visit and be given the option to participate in an open-label rollover extension and receive bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) until it becomes commercially available, or until Gilead Sciences elects to terminate the development of BIC/F/TAF.
  Interventions: Drug: BIC; Drug: F/TAF; Drug: DTG Placebo; Drug: B/F/TAF
- DTG + F/TAF (Active Comparator): Participants will receive DTG + F/TAF FDC + BIC placebo for 48 weeks.
  * Following Week 48, participants will continue to take their blinded treatment and attend visits every 12 weeks until treatment assignments have been unblinded. Participants will return for an unblinding visit and be given the option to participate in an open-label rollover extension and receive B/F/TAF until it becomes commercially available, or until Gilead Sciences elects to terminate the development of BIC/F/TAF.
  Interventions: Drug: F/TAF; Drug: DTG; Drug: BIC Placebo; Drug: B/F/TAF
- Open Label Extension Phase (Experimental): After Week 48 participants continued to take their randomized study drug and attended visits every 12 weeks until treatment assignments were unblinded, at which point all participants returned for an unblinding visit and were given the option to participate in an open-label rollover extension to receive an FDC containing B/F/TAF.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: BIC — 75 mg tablet administered orally once daily
  Other Names: GS-9883
  Arms: BIC + F/TAF
Drug: F/TAF — 200/25 mg FDC tablet administered orally once daily
  Arms: BIC + F/TAF; DTG + F/TAF
Drug: DTG — 50 mg tablet administered orally once daily
  Other Names: Tivicay®
  Arms: DTG + F/TAF
Drug: BIC Placebo — Tablet administered orally once daily
  Arms: DTG + F/TAF
Drug: DTG Placebo — Tablet administered orally once daily
  Arms: BIC + F/TAF
Drug: B/F/TAF — 50/200/25 mg FDC tablet administered orally once daily

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of bictegravir (BIC) + emtricitabine/tenofovir alafenamide (F/TAF) fixed dose combination (FDC) versus dolutegravir (DTG) + F/TAF in HIV-1 Infected, antiretroviral treatment-naive adults. This study will also evaluate the pharmacokinetic (PK) profile of BIC, emtricitabine and TAF.

ELIGIBILITY:
Key Inclusion Criteria:

* Antiretroviral naive (≤ 10 days of prior therapy with any antiretroviral agent)
* Plasma HIV-1 RNA levels ≥ 1,000 copies/mL at screening
* Screening genotype report provided by Gilead Sciences must show sensitivity to tenofovir (TFV) and emtricitabine (FTC)
* Adequate renal function as measured by estimated glomerular filtration rate ≥ 70 mL/min according to the Cockcroft-Gault formula
* CD4+ cell count ≥ 200 cells/µL at screening

Key Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to screening as defined in the study protocol
* Prior use of antiretrovirals in the setting of pre-exposure prophylaxis (PrEP) or post exposure prophylaxis (PEP)
* Chronic hepatitis B virus (HBV) infection
* Hepatitis C infection (Individuals who are hepatitis C virus (HCV) Ab positive, but have a documented negative HCV RNA, are eligible)
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Participation in any other clinical trial without prior approval from the sponsor is prohibited while participating in this trial

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (18):
- United States (18):
  - Phoenix, Arizona
  - Los Angeles, California
  - Sacramento, California
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Boston, Massachusetts
  - Berkley, Michigan
  - Newark, New Jersey
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Longview, Texas
  - Annandale, Virginia
  - Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sax PE, DeJesus E, Crofoot G, Ward D, Benson P, Dretler R, Mills A, Brinson C, Peloquin J, Wei X, White K, Cheng A, Martin H, Quirk E. Bictegravir versus dolutegravir, each with emtricitabine and tenofovir alafenamide, for initial treatment of HIV-1 infection: a randomised, double-blind, phase 2 trial. Lancet HIV. 2017 Apr;4(4):e154-e160. doi: 10.1016/S2352-3018(17)30016-4. Epub 2017 Feb 15. PMID 28219610
- [Result] Sax PE, DeJesus E, Crofoot G, Ward D, Benson P, Dretler R, Mills A, Brinson C, Wei X, Collins SE, Cheng A. Coformulated bictegravir, emtricitabine, tenofovir alafenamide after initial treatment with bictegravir or dolutegravir and emtricitabine/tenofovir alafenamide. AIDS. 2018 Jul 31;32(12):1723-1725. doi: 10.1097/QAD.0000000000001894. PMID 29794828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 22 centers in the United States of America.The first participant was screened on 23 March 2015 and the last study visit occurred on 27 February 2019.
Pre-assignment Details: 125 participants were screened.
Groups:
- BIC + F/TAF: Bictegravir (BIC) (75 mg) + emtricitabine/tenofovir alafenamide (F/TAF) (200/25 mg) fixed-dose combination (FDC) + dolutegravir (DTG) placebo tablets orally once daily for 48 weeks. After Week 48 participants continued to take their randomized study drug and attended visits every 12 weeks until treatment assignments were unblinded, at which point all participants returned for an unblinding visit and were given the option to participate in an open-label rollover extension to receive an FDC containing B/F/TAF (50/200/25 mg).
- DTG + F/TAF: DTG (50 mg) + F/TAF (200/25 mg) FDC + BIC placebo tablets orally once daily. After Week 48 participants continued to take their randomized study drug and attended visits every 12 weeks until treatment assignments were unblinded, at which point all participants returned for an unblinding visit and were given the option to participate in an open-label rollover extension to receive an FDC containing B/F/TAF (50/200/25 mg).
Period: Double-Blinded Phase
Arm/Group | BIC + F/TAF | DTG + F/TAF
Started | 65 | 33
Completed | 62 | 30
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Non-compliance with study drug | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Period: Open Label Extension Phase
Arm/Group | BIC + F/TAF | DTG + F/TAF
Started | 62 | 30
Completed | 54 | 29
Not Completed | 8 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrew Consent | 3 | 1
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- BIC + F/TAF: BIC 75 mg + F/TAF (200/25 mg) FDC + DTG placebo tablets orally once daily for 48 weeks. After Week 48 participants continued to take their randomized study drug and attended visits every 12 weeks until treatment assignments were unblinded, at which point all participants returned for an unblinding visit and were given the option to participate in an open-label rollover extension to receive an FDC containing B/F/TAF (50/200/25 mg).
- DTG + F/TAF: DTG 50 mg + F/TAF (200/25 mg) FDC + BIC placebo tablets orally once daily. After Week 48 participants continued to take their randomized study drug and attended visits every 12 weeks until treatment assignments were unblinded, at which point all participants returned for an unblinding visit and were given the option to participate in an open-label rollover extension to receive an FDC containing B/F/TAF (200/50/25 mg).
- Total: Total of all reporting groups
Arm/Group | BIC + F/TAF | DTG + F/TAF | Total
Number analyzed (Participants) | 65 | 33 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11.4) | 38 (12.9) | 35 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 64 | 30 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Black | 24 | 12 | 36
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
  White | 38 | 18 | 56
  Other | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 4 | 15
  Not Hispanic or Latino | 54 | 29 | 83
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.39 (0.764) | 4.38 (0.866) | 4.39 (0.795)
HIV-1 RNA category [Count of Participants; unit: Participants]
  ≤ 100,000 copies/mL | 55 | 26 | 81
  > 100,000 to ≤ 400,000 copies/mL | 6 | 6 | 12
  > 400,000 copies/mL | 4 | 1 | 5
CD4 Cell Count [Mean (Standard Deviation); unit: cells/μL] | 471 (190.9) | 507 (271.0) | 483 (220.3)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  < 200 cells/μL | 3 | 3 | 6
  ≥ 200 to < 350 cells/µL | 17 | 8 | 25
  ≥ 350 to < 500 cells/µL | 20 | 6 | 26
  ≥ 500 cells/µL | 25 | 16 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL as Determined by the FDA-defined Snapshot Algorithm.
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Full Analysis Set included all participants who were randomized into the double-blinded phase of study and received at least 1 dose of study drug during the double-blinded phase.
Measure: Number; unit: percentage of participants
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 65 | 33
percentage of participants | 96.9 | 93.9
Statistical Analysis 1: Comparison: BIC + F/TAF vs DTG + F/TAF; Test type: Non-Inferiority — Noninferiority of treatment with BIC + F/TAF relative to treatment with DTG + F/TAF. Noninferiority assessed using a conventional 95% confidence interval (CI) approach, with a noninferiority margin of 12%; p = 0.5, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel test stratified by baseline HIV-1 RNA stratum (≤ 100,000 copies/mL vs > 100,000 copies/mL); Difference in percentages = 2.9, 95% CI 2-sided [-8.5 to 14.2]

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL as Determined by the FDA-defined Snapshot Algorithm at Week 12
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 12 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 65 | 33
percentage of participants | 93.8 | 93.9

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL as Determined by the FDA-defined Snapshot Algorithm at Week 48
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 65 | 33
percentage of participants | 96.9 | 90.9

4. Secondary Outcome: The Change From Baseline in log10 HIV-1 RNA at Week 12
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 64 | 31
log10 copies/mL | -3.03 (0.791) | -3.15 (0.731)

5. Secondary Outcome: The Change From Baseline in log10 HIV-1 RNA at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 64 | 32
log10 copies/mL | -3.09 (0.740) | -3.12 (0.757)

6. Secondary Outcome: The Change From Baseline in log10 HIV-1 RNA at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 63 | 32
log10 copies/mL | -3.09 (0.752) | -3.11 (0.852)

7. Secondary Outcome: The Change From Baseline in Cluster of Differentiation 4 Positive (CD4+) Cell Count at Week 12
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: CD4 Cell Count (/μL)
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 64 | 31
CD4 Cell Count (/μL) | 170 (150.0) | 173 (220.5)

8. Secondary Outcome: The Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: CD4 Cell Count (/μL)
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 64 | 32
CD4 Cell Count (/μL) | 190 (176.8) | 155 (165.8)

9. Secondary Outcome: The Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: CD4 Cell Count (/μL)
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 63 | 30
CD4 Cell Count (/μL) | 258 (221.7) | 188 (238.7)

10. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) During Double-Blinded Randomized Phase
Time Frame: First dose date up to last dose (maximum duration: 58 Weeks) plus 30 days (During Double-Blinded Randomized Phase)
Population: Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- BIC + F/TAF: BIC 75 mg + F/TAF (200/25 mg) FDC + DTG placebo tablets orally once daily for 48 weeks. After Week 48 participants continued to take the study drug and attended visits every 12 weeks until treatment assignments were unblinded, at which point all participants returned for an unblinding visit and were given the option to participate in an open-label rollover extension to receive an FDC containing B/F/TAF (50/200/25 mg).
- DTG + F/TAF: After participants completed their blinded treatment with DTG 50 mg + F/TAF 200/25 mg FDC + BIC placebo, they were given the option to participate in an open-label rollover extension to receive an FDC containing B/F/TAF (200/50/25).
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 65 | 33
percentage of participants | 87.7 | 72.7

11. Secondary Outcome: Percentage of Participants With Treatment Emergent Laboratory Abnormalities During Double-Blind Randomized Phase
Time Frame: First dose date up to last dose (maximum duration: 58 Weeks) plus 30 days (During Double-Blinded Randomized Phase)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 65 | 33
percentage of participants | 87.5 | 87.5

12. Secondary Outcome: PK Parameter: Cmax for Bictegravir (BIC), Emtricitabine (FTC), Tenofovir Alafenamide (TAF) and Tenofavir (TFV) at Steady-State
Description: Cmax is the maximum observed plasma concentration of the drug.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Week 4 or 8
Population: Pharmacokinetic (PK) Substudy Analysis Set included all participants who (1) were randomized into the double-blinded phase of study, (2) were enrolled into the PK substudy, (3) received at least 1 dose of study drug during the double-blinded phase, and (4) had at least 1 nonmissing intensive PK concentration value.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 23 | 7
ng/mL
  BIC | 9344.3 (2506.33) | NA (NA) — Participants did not receive BIC
  FTC: number analyzed (Participants) | 22 | 7
  FTC | 1919.1 (470.18) | 2157.1 (486.44)
  TAF | 249.1 (137.40) | 260.8 (212.44)
  TFV | 19.1 (4.50) | 20.9 (8.16)

13. Secondary Outcome: PK Parameter: Tmax for BIC, FTC, TAF, and TFV at Steady-State
Description: Tmax was defined as the time to Cmax.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Week 4 or 8
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 23 | 7
hours
  BIC | 2.00 [1.50 to 3.00] | NA [NA to NA] — Participants did not receive BIC
  FTC | 1.50 [1.00 to 2.00] | 1.50 [1.02 to 2.00]
  TAF | 1.00 [0.50 to 1.50] | 1.00 [0.50 to 1.00]
  TFV | 1.50 [1.50 to 2.00] | 2.00 [1.53 to 2.00]

14. Secondary Outcome: PK Parameter:Ctau for BIC, FTC and TFV
Description: Ctau was defined as the observed drug concentration at the end of the dosing interval.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Week 4 or 8
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 23 | 7
ng/mL
  BIC | 3508.6 (1288.85) | NA (NA) — Participants did not receive BIC
  FTC | 76.6 (26.35) | 102.6 (57.60)
  TFV | 10.7 (2.65) | 12.2 (5.02)

15. Secondary Outcome: PK Parameter: AUCtau for BIC, FTC, TAF, and TFV
Description: AUCtau is defined as the area under the concentration-time curve of the drug over time.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Week 4 or 8
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 23 | 7
h*ng/mL
  BIC | 139778.8 (37810.07) | NA (NA) — Participants did not receive BIC
  FTC | 11605.4 (3241.84) | 14689.8 (5869.37)
  TAF | 247.4 (140.62) | 245.6 (125.03)
  TFV | 316.0 (74.01) | 369.4 (147.96)

16. Secondary Outcome: PK Parameter: t1/2 of BIC, FTC, TAF, and TFV
Description: t1/2 was defined as the terminal elimination half-life of the drug
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours postdose at Week 4 or 8
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | BIC + F/TAF | DTG + F/TAF
Number analyzed (Participants) | 23 | 7
hours
  BIC | 16.73 [13.79 to 19.28] | NA [NA to NA] — Participants did not receive BIC
  FTC | 5.46 [5.19 to 6.11] | 5.70 [5.3 to 6.38]
  TAF | 0.37 [0.28 to 0.49] | 0.42 [0.40 to 0.45]
  TFV | 37.74 [28.26 to 48.40] | 34.47 [31.97 to 47.57]

ADVERSE EVENTS:
Time Frame: First dose date to last dose date of BIC + F/TAF or B/F/TAF (maximum duration: 193.4 weeks) plus 30 days
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- BIC + F/TAF (Double-Blind Randomized): Adverse events in this reporting group include those that occurred during the double-blind phase by participants randomized to BIC + F/TAF. Participants received BIC (75 mg) + F/TAF (200/25 mg) FDC + DTG placebo tablets orally once daily for 48 weeks.
- DTG + F/TAF (Double Blind Randomized):: Adverse events in this reporting group include those that occurred during the double-blind phase by participants randomized to DTG + FTC/TAF. Participants received DTG (50 mg) + F/TAF (200/25 mg) FDC + BIC placebo tablets orally once daily.
- BIC + F/TAF to B/F/TAF (Open-Label Phase): Adverse events reported occurred during the Open-Label Extension Phase in participants who enrolled into the Extension Phase from the BIC + F/TAF group and received B/F/TAF (50/200/25 mg) FDC tablet.
- DTG + F/TAF to B/F/TAF (Open-Label Phase): Adverse events reported occurred during the Open-Label Extension Phase in participants who enrolled into the Extension Phase from the DTG + F/TAF group and received B/F/TAF (50/200/25 mg) FDC tablet.
Arm/Group | BIC + F/TAF (Double-Blind Randomized) | DTG + F/TAF (Double Blind Randomized): | BIC + F/TAF to B/F/TAF (Open-Label Phase) | DTG + F/TAF to B/F/TAF (Open-Label Phase)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/33 | 0/62 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/65 | 0/33 | 3/62 | 5/30
Other Adverse Events (participants affected / at risk) | 44/65 | 18/33 | 42/62 | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIC + F/TAF (Double-Blind Randomized) (N=65) | DTG + F/TAF (Double Blind Randomized): (N=33) | BIC + F/TAF to B/F/TAF (Open-Label Phase) (N=62) | DTG + F/TAF to B/F/TAF (Open-Label Phase) (N=30)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Bladder mass (Renal and urinary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIC + F/TAF (Double-Blind Randomized) (N=65) | DTG + F/TAF (Double Blind Randomized): (N=33) | BIC + F/TAF to B/F/TAF (Open-Label Phase) (N=62) | DTG + F/TAF to B/F/TAF (Open-Label Phase) (N=30)
Anal fissure (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 4 | 4 | 4
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 3 | 2 | 3
Chest pain (General disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 3 | 0
Pain (General disorders) | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 2 | 3
Chlamydial infection (Infections and infestations) | 4 | 2 | 4 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 2
Furuncle (Infections and infestations) | 3 | 2 | 4 | 2
Gastroenteritis (Infections and infestations) | 1 | 2 | 1 | 2
Gonorrhoea (Infections and infestations) | 3 | 1 | 5 | 2
Influenza (Infections and infestations) | 1 | 1 | 4 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1 | 3 | 3
Pharyngitis (Infections and infestations) | 2 | 1 | 3 | 2
Proctitis gonococcal (Infections and infestations) | 1 | 1 | 2 | 5
Sinusitis (Infections and infestations) | 3 | 0 | 4 | 2
Syphilis (Infections and infestations) | 3 | 1 | 8 | 5
Upper respiratory tract infection (Infections and infestations) | 7 | 1 | 4 | 1
Urethritis (Infections and infestations) | 3 | 3 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2
Viral infection (Infections and infestations) | 0 | 2 | 2 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 2 | 2 | 6 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 5 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 6 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 1
Stress (Psychiatric disorders) | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 7 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years